CLINICAL TRIAL: NCT00205322
Title: A Phase II Study of Oxaliplatin, 5-fluorouracil, and Leucovorin in Combination With Oral Capecitabine in Patients With Metastatic Colorectal Cancer
Brief Title: Oxaliplatin, 5-FU and Leucovorin in Combination With Oral Capecitabine for Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO03216; M-2003-0544 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH/MEDICINE/H (Other: UW Madison)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2011-12

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy; Capecitabine; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: chemotherapy (capecitabine, oxaliplatin, 5-FU, leucovorin)

SUMMARY:
The combination of oxaliplatin, 5-FU, leucovorin, and capecitabine is hypothesized to retain and potentially improve upon the activity of the FOLFOX regimens. Additionally, the use of an oral rather than an infusional 5-fu regimen represents a clear advantage in terms of both patient convenience and lack of associated catheter-related complications.

ELIGIBILITY:
Inclusion Criteria:

* no prior treatment for metastatic disease
* PS 0-2
* measurable disease

Exclusion Criteria:

* neuropathy > or equal to grade 2
* concomitant radiation therapy or other systemic cancer therapies
* brain mets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Does the combination of oxaliplatin, 5-FU, leucovorin and capecitabine improve the activity of the FOLFOX regimens in metastatic colorectal cancer patients | Bi-monthly collection of information regarding tumor progression and overall survival.

SECONDARY OUTCOMES:
Is the oral drug an advantage in this patient population | Bi-monthly collection of information regarding tumor progression and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mulkerin, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu